CLINICAL TRIAL: NCT03411642
Title: Comparative Effectiveness Study of Transthoracic and Transesophageal Echocardiography in Stroke
Acronym: CONTEST
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Albertinen Krankenhaus (Other); Regio Kliniken (Other); Helios University Hospital Wuppertal (Other); Kreiskliniken Reutlingen (Other); Klinikum Karlsbad-Langensteinbach (Other)
Responsible Party: Sponsor
Other Study IDs: PV5225
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Acute
Keywords: Stroke, echocardiography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Comparative Effectiveness Study of Transthoracic and Transesophageal Echocardiography in Stroke (CONTEST) aims at assessing the diagnostic value of transesophageal echocardiography (TEE) and transthoracic echocardiography (TTE) with regards to treatment consequences in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
For this purpose, the investigators will perform a prospective multicenter diagnostic comparative effectiveness study. Patients with acute stroke will be studied by both TTE and TEE. Patients with already defined stroke etiology and determined secondary prevention will be excluded from the trial. Treatment relevant diagnostic findings will be identified by a central endpoint adjudication committee. In order to demonstrate a hypothesized 2% absolute increase in the number of treatment relevant diagnostic findings by TEE as compared to TTE, 880 stroke patients will be enrolled in six German stroke centers. CONTEST will allow answering the question whether and for which group of stroke patients TEE is indicated in addition to TTE. By this, the study will provide evidence to guide justified recommendations for echocardiography in acute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke or transitory ischemic attack (TIA)
* age ≥18 years
* informed consent

Exclusion Criteria:

* Patients with already defined stroke etiology and determined secondary prevention treatment strategy prior to echocardiography (e.g. atrial fibrillation, carotid artery stenosis, cervical artery dissection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute stroke in whom echocardiography is indicated will be studied by TTE and TEE.
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Götz Thomalla, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (4):
- Germany (4):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Albertinen-Krankenhaus, Hamburg
  - Regio Klinikum Pinneberg, Pinneberg
  - Kreiskliniken Reutlingen, Reutlingen

REFERENCES:
- [Derived] Thomalla G, Upneja M, Camen S, Jensen M, Schroder J, Barow E, Boskamp S, Ostermeier B, Kissling S, Leinisch E, Tiburtius C, Clausen H, Cheng B, Blankenberg S, Nedelmann M, Steinbrecher A, Andres F, Rosenkranz M, Sinning C, Schnabel RB, Gerloff C. Treatment-Relevant Findings in Transesophageal Echocardiography After Stroke: A Prospective Multicenter Cohort Study. Stroke. 2022 Jan;53(1):177-184. doi: 10.1161/STROKEAHA.121.034868. Epub 2021 Sep 9. PMID 34496617

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Included: All patients with acute ischemic stroke and undetermined origin at study inclusion who were enrolled and planned to be studied with both TTE and TEE
Period: Overall Study
Arm/Group | Patients Included
Started | 494
Participants Who Received TTE | 492
Participants Who Received TEE | 454
Completed | 454 (454 patients received both TEE and TTE)
Not Completed | 40

BASELINE CHARACTERISTICS:
Arm/Group | Patients Included
Number analyzed (Participants) | 494
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204
  Male | 290
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 494
Diagnosis (acute ischemic stroke, transient ischemic attack, retinal ischemia) [Count of Participants; unit: Participants]
  Acute ischemic stroke | 385
  Transient ischemic attack | 89
  Retinal ischemia | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Diagnostic Findings That Lead to a Change in Acute Treatment or Treatment for Secondary Prevention
Description: Treatment relevant diagnostic findings identified by a central endpoint adjudication committee comprising both cardiologists and neurologists.
Time Frame: Inpatient treatment on a stroke unit usually <7 days
Measure: Count of Participants; unit: Participants
Groups:
- Patients Studied With Both TTE and TEE: Patients studied with both TTE and TEE
Arm/Group | Patients Studied With Both TTE and TEE
Number analyzed (Participants) | 454
Participants
  Treatment relevant findings in TTE: Yes | 64
  Treatment relevant findings in TTE: No | 390
  Treatment relevant findings in TEE: Yes | 86
  Treatment relevant findings in TEE: No | 368

2. Secondary Outcome: Number of Patients With Change of Assessment of Stroke Etiology After TEE
Description: Number of patients with change in the assessment of stroke etiology (cardioembolism, large artery atherosclerosis, small vessel disease, other determined etiology, unknown etiology) after performing TEE
Time Frame: Inpatient treatment on a stroke unit usually <7 days
Population: All patients studied with TTE and TEE
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Studied With Both TTE and TEE
Number analyzed (Participants) | 454
Participants
  Yes | 52
  No | 401
  Missing data | 1

ADVERSE EVENTS:
Time Frame: In-patient treatment on a stroke unit usually <7 days
Description: Investigator recorded all events considered related to TTE or TEE
Groups:
- Patients Receiving TTE: All patients with acute ischemic stroke and undetermined origin at study inclusion who were enrolled studied with TTE
- Patients Receiving TEE: All patients with acute ischemic stroke and undetermined origin at study inclusion who were enrolled studied with TEE
Arm/Group | Patients Receiving TTE | Patients Receiving TEE
All-Cause Mortality (participants affected / at risk) | 0/492 | 0/454
Serious Adverse Events (participants affected / at risk) | 0/492 | 0/454
Other Adverse Events (participants affected / at risk) | 0/492 | 0/454

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03411642/Prot_SAP_000.pdf